CLINICAL TRIAL: NCT00385463
Title: A Multicenter, Randomized, Double-Blind, Triple-Dummy, Placebo-Controlled, Parallel Group, Four-Week Study Assessing the Efficacy of Fluticasone Propionate Aqueous Nasal Spray Versus Montelukast in Adolescents/Adults With Asthma and Seasonal Allergic Rhinitis Receiving Advair Diskus(R) or Placebo
Brief Title: Adolescent and Adult Subjects With Asthma and Seasonal Allergic Rhinitis Receiving Advair Diskus or Placebo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSK ADA103575
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Asthma; Seasonal Allergic Rhinitis
Keywords: Asthma; Rhinitis; Allergic Asthma
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Seasonal; Rhinitis | interventions — BID protein, human; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Adding Advair Diskus 100/50mcg (FSC) BID and Singulair 10mg is added to placebo Diskus BID

SUMMARY:
The four respiratory drugs being researched in this study have been approved by the US Food and Drug Administration (FDA) and are currently available by prescription at your drug store. One of the drugs is for the treatment of asthma alone, one is for treatment of SAR alone, and one is for treatment of both SAR and asthma. In addition, you will also receive one asthma rescue drug (albuterol) that is to be used for any breakthrough asthma symptoms that you may experience throughout the study.

The purpose of this study is to see how well your asthma and SAR are controlled when taking one of the medicine combinations

DETAILED DESCRIPTION:
4-week study to assess asthma control as measured by lung function and clinical features, rhinitis treatment, subject-rated overall satisfaction with treatment, and safety outcomes when FLONASE™ 200mcg (FPANS) QD, Singulair 10mg (MON) QD, or placebo QD is added to ADVAIR™ DISKUS™ 100/50mcg (FSC) BID and when Singulair 10mg (MON) QD is added to placebo DISKUS BID in adolescent and adults subjects. Male or female subjects must be symptomatic with both seasonal allergic rhinitis and persistent asthma, and have an FEV1 65-95% of predicted while using an as-needed short-acting beta2-agonist or an allowed ICS or non-ICS controller therapy. Subjects will replace their short-acting beta2-agonist with VENTOLIN™ HFA (for rescue) and will enter a 7-14 day run-in period during which they will continue use of their pre-study controller therapy. At Visit 2, subjects who meet both the asthma and rhinitis randomization criteria will be randomized to double-blind treatment with ADVAIR DISKUS 100/50mcg BID and either FLONASE 200mcg QD, Singulair 10mg QD, or placebo QD, or to placebo DISKUS BID and Singulair 10mg QD. The co-primary efficacy measures will be the mean change from baseline at endpoint in AM PEF, compared between the FSC and the MON treatment groups to assess superiority and compared between the FSC and FSC+MON treatment groups to assess equivalence. Secondary efficacy measures for rhinitis will be mean change from baseline in subject-rated daytime total nasal symptom score and nighttime total nasal symptomatic score averaged over Weeks 1-2 (D-TNSSW1-2 and N-TNSSW1-2, respectively). Secondary efficacy measures for asthma will be mean change from baseline at endpoint in morning pre-dose FEV1, percentage of symptom-free days, and percentage of rescue-free days. Other measures will include subject-rated overall satisfaction with treatment, evening PEF, asthma symptom scores (D-INSSW1-x, N-INSSW1-2), averaged over Weeks 1-2. Descriptive measures will include all total and individual nasal symptoms scores averaged over Weeks1-4. Safety measures will include assessment of clinical adverse events and asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent is obtained.
* Male or female
* 15 Years and older
* Diagnosis of persistent asthma for at least three months.
* 3 months prior and current use of specified asthma therapies
* FEV1 between 65-95% of predicted value
* Diagnosis of seasonal allergic rhinitis
* Active residence within geographical regions where exposure to relevant seasonal allergic is expected

Exclusion Criteria:

* Currently diagnosed with life-threatening asthma
* Asthma instability
* Concurrent respiratory disease
* Nasal obstruction
* Nasal history
* Certain concurrent conditions/diseases
* Drug allergy
* Respiratory tract infections
* Specific (listed in protocol) concurrent medications
* Systemic corticosteroids

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline at endpoint in morning PEF compared between fluticasone propionate/salmeterol combination product 100/50mcg BID (FSC) and montelukast 10mg QD (MON) treatment groups.
Assess superiority and compare between FSC and FSC+MON treatment groups
Assess equivalence.

SECONDARY OUTCOMES:
Rhinitis mean change from baseline in subject-rated: daily, total nasal symptom scores averaged over Weeks 1-2 and nighttime total nasal symptom scores averaged over Weeks 1-2.
Asthma assess superiority and assess equivalence: mean change from baseline at endpoint in predose AM FEV1; percentage of asthma rescue-free days; and percentage of asthma rescue-free days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Townley, M.D., Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States